CLINICAL TRIAL: NCT06599489
Title: Sleeve Gastrectomy With Crural Repair With or Without Ligamentum Teres Wrapping in Obese Patients With Gastroesophageal Reflux Disease .Arandomized Controlled Trial
Brief Title: Management of Obese Patients With Gastroesophageal Reflux Disease .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hossam Mahmoud Ibrahim (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Hossam Mahmoud Ibrahim, Assistant lecturer at general surgery department, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: obesity and GERD
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity and reflux
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux | interventions — Heller Myotomy

STUDY DESIGN:
Intervention Model Description: operation surgical intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeve gastrectomy and cruroplasty (Other): Under a general anesthesia. Three 12-mm trocars were inserted in the upper abdomen and one 5-mm trocar was inserted laterally in the left-upper quad¬rant. Retractor was inserted through the subxyphoid 10 mm trocar site to re¬tract the liver (five to seven Trocars always used) . The hiatal hernia sac containing the proximal stomach was reduced. Distal esophagus and gastroesophageal junction were mobilized by using a laparoscopic Harmon¬ic Scalpelto get a 4-cm tension-free intra-abdominal esophagus. Pos¬terior crural repair was performed with three interrupt¬ed
  Interventions: Procedure: surgery ..operation
- sleeve gastrectomy and cruroplasty with ligamentum teres wrapping (Other): sleeve gastrectomy and cruroplasty with ligamentum teres wrapping for cardiopexy for morbidly obese patients with reflux symptomspatients will Laparoscopic sleeve gastrectomy with crural repair with ligamentum teres wrapping .the same as in group (A) in addition to ligamentum teres wrapping behind lower end of oesophagus and fixed to anterior wall of stomach with interrupted sutures .
  The mean follow up period was eight months .clinical outcomes were also evaluated in term of GERD symptoms improvement or resolution .interruption of anti reflux medications and xray evidence of HH recurrence.
  Interventions: Procedure: surgery ..operation

INTERVENTIONS:
Procedure: surgery ..operation — sleeve gastrectomy with cruroplasty with or without ligamentum teres wrapping
  Other Names: sleeve gastrectomy and cruroplasty; ligamentum teres wrapping

SUMMARY:
The aim of this study is to evaluate the efficacy Sleeve gastrectomy with cruroplasty with or without ligamentum teres wrapping for management of morbidly obese patients with concomitant reflux symptoms.

DETAILED DESCRIPTION:
All patients underwent a preoperative work-up including history and physical examination, routine laboratory investigations, ECG, chest radiography, pulmonary function tests, abdominal ultrasonography, and barium swallow, upper GIT endos¬copy, 24 hours PH monitoring, nutritional, and psychiat¬ric evaluation. Further exams and/or consultations were performed when indicated. The study design was a pro¬spective randomized controlled study that received ap¬proval from the ethics committee in relevant hospitals. All the patients gave an informed written consent All patients had a written informed consent of the two types laparoscopic procedures of obesity, Prophylactic anticoagulant medications will be given to all patients in the form of subcutaneous Clexane 0.5 unit/Kg/24. An Intensive care unit (ICU) bed will be reserved for all patients the night of operation with the decision of transfer left to the postoperative recovery assessment.

According to the patient selection, all patients will be divided into two groups as follows:

Group (A): Patients will do Laparoscopic sleeve gastrectomy with crural repair. Under a general anesthesia, the patient was placed in the split-leg position with the surgeon standing between the legs and the assistant on the left-hand side of the pa¬tient. A veress needle was used to create the pneumoperi-toneum. Three 12-mm trocars were inserted in the upper abdomen (one on the right, two on the left side) and one 5-mm trocar was inserted laterally in the left-upper quad¬rant. Retractor was inserted through the subxyphoid 10 mm trocar site to re¬tract the liver (five to seven Trocars always used) The hiatal hernia sac containing the proximal stomach was reduced. Distal esophagus and gastroesophageal junction were mobilized by using a laparoscopic Harmon¬ic Scalpel (Ethicon Endo-Surgery Inc., Cincinnati, OH) to get a 4-cm tension-free intra-abdominal esophagus. Pos¬terior crural

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* Both sexes.
* BMI ≥ 40 or ≥ 35 with co-morbidity.with reflux symptoms .
* Failure of non-surgical treatment.
* Patients with hiatus hernia .
* Absence of endocrinal or psychological disorders.
* Failure of non surgical treatment
* Non sweat eaters
* Patients with no previous upper GIT surgeries

Exclusion Criteria:

* Presence of endocrinal or psychological disorders.
* Morbidly obese patients with no reflux symptoms
* sweat eaters
* Patients with barrett,s oesophagus ,
* Patient with bad general condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss and improvement of BMI | 6 momths
  BMI from above 35 kg/m2 to less,than 30. kg /m2to be less than 35 kg /m2
Reflux symptoms | 6 months
  Improvement of all symptoms of reflux disease

CONTACTS AND LOCATIONS:
Overall Officials: Assiut university, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No